CLINICAL TRIAL: NCT03132181
Title: Empagliflozin as a Modulator of Systemic Vascular Resistance and Cardiac Output in Patients With Type 2 Diabetes
Acronym: EMPA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: RWTH Aachen University (Other)
Collaborators: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 15-124
Record Dates: First submitted 2017-04-20; First posted 2017-04-27 (Actual); Last update posted 2019-02-12 (Actual); Status verified 2019-02

CONDITIONS: Diabetes Mellitus Type 2 (T2DM)
Keywords: Empagliflozin; Diabetes; Systemic vascular resistance; Cardiac output; Blood pressure
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — empagliflozin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Empagliofizin (Experimental): Patients will receive empagliflozin 10 mg qd for a period of 3 months.
  Interventions: Drug: Empagliflozin
- Placebo (Placebo Comparator): Patients of the placebo arm will receive placebo tablets qd for a period of 3 months.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Empagliflozin — Patient will be treaded according to standard care but additionally take one tablet Empagliflozin per day
  Other Names: Jardiance
  Arms: Empagliofizin
Other: Placebo — Patient will be treaded according to standard care but additionally take one tablet placebo per day
  Arms: Placebo

SUMMARY:
SGLT2 inhibitors are a novel class of glucose lowering drugs that act in the kidney by inhibiting SGLT2-mediated glucose reabsorption in the proximal tubule. The resulting increase in urinary glucose excretion leads to a reduction in plasma glucose levels. This is accompanied by reduction of total body weight due to urinary energy loss. In addition, glucose dependent osmotic diuresis contributes to blood pressure lowering effects of SGLT2 inhibition.

Aim of the trial is to assess hemodynamic changes by empagliflozin, identify new empagliflozin dependent metabolic regulators and evaluate empagliflozin dependent effects on cardiac function.

DETAILED DESCRIPTION:
Strikingly, empagliflozin was recently found to reduce cardiovascular mortality in addition to heart failure in the EMPA-REG OUTCOME trail. This multi-center, randomized, placebo controlled study enrolled 7020 patients with type 2 diabetes at high cardiovascular risk. Patients were randomized to placebo or one of 2 doses of empagliflozin (10 or 25 mg/d) on the background of state-of-the-art glucose-lowering therapy with good control of associated CV risk factors at trial entry. At the end of the study, empagliflozin led to a slightly lower HbA1c of 0.3 - 0.4 % in comparison to placebo with higher addition of other anti-hyperglycemic medications found in the placebo group. Moreover, empagliflozin compared with placebo led to a significant reduction in blood pressure and body weight, similar to what has been reported in earlier studies. For the primary outcome empagliflozin significantly reduced the risk of cardiovascular death, myocardial infarction and stroke compared with placebo with a hazard ratio of 0.86 (95% CI 0.74-0.99; p=0.038). This reduction was mainly driven by a highly significant 38% reduction in cardiovascular death (HR 0.62; 95% CI 0.49-0.77), with a very early separation of the curves evident as early as 2 months into the trial. There was a non-significant 13% reduction of non-fatal myocardial infarction (p=0.30) and a non-significant 24% increased risk for non-fatal stroke (p=0.16). In addition, in a secondary/exploratory analysis, empagliflozin led to a significant reduction of hospitalization for heart failure with a 35% risk reduction (HR 0.65; 95% CI 0.50-0.85; p<0.002), with separation of the curves evident almost immediately during trial observation, suggesting a very early effect of the SGLT2-inhibitor. Finally, empagliflozin reduced overall mortality by 32% (HR 0.68; 95% CI 0.57-0.82; p<0.0001), a highly significant effect translating into a number-needed-to-treat (NNT) of 39 over 3 years to prevent one death.

These large unexpected, beneficial effects of empagliflozin on all-cause death, CV death and HF hospitalization have raised important questions, as to the mechanism underpinning these favorable CV actions, which cannot be explained by glucose control nor a reduction of atherosclerotic events.

The rapid separation of survival and HF-event curves suggest an instant mode of empagliflozin action - which we here hypothesize to be driven by immediate changes of hemodynamic parameters. This might be followed by more delayed metabolic effects contributing to the beneficial risk profile.

The investigators speculate empagliflozin dependent hemodynamic changes to be responsible for the early and longer term blood pressure lowering effects. This might initially be driven a rapidly occurring empagliflozin dependent natriuresis.

This hypothesis is based on:

* The glucosuric effects of SGLT2 inhibitors leading - at least temporarily- to an increase in sodium excretion as well as a reduction in plasma volume due to glucose osmotic diuretic effects and natriuresis
* SGLT2 inhibition has been suggested to directly affect the tubulo-glomerular feedback mechanism in the kidney. The increased delivery of solute (sodium and chloride) to the macula densa in the setting of SGLT2 inhibition may reduce hyperglycemia-induced glomerular hyperfiltration via tubulo-glomerular feedback invoking adenosine-dependent pathways, with direct effects on afferent glomerular arteriolar tone that may diminish hyperfiltration acutely and consistently during treatment. Moreover, these hemodynamic effects may possibly lead to aldosterone withdrawal (thus mimicking to some degree the efficacy of mineralocorticoid antagonism) as well as contributing to inhibition of sympathetic activation.
* Several trials have shown that SGLT2-inhibitors lead to a reduction in systolic blood pressure in a range of 3-5 mmHg and about 2-3 mmHg in diastolic blood pressure. In addition, SGLT2-inhibitors reduce pulse pressure, mean arterial pressure and the product of heart rate-X-systolic blood pressure (a.k.a. "double product") vs. placebo suggesting an effect on different markers and mediators of arterial stiffness. Interestingly, these BP effects occurred without a compensatory increase in heart rate, suggesting a lack of compensatory sympathetic activation. Various mechanisms may contribute to the reduction in BP including weight loss, diuretic effects (osmotic diuresis and natriuresis), sodium depletion but also potential direct and indirect effects on arteriolar relaxation and oxidative stress. In a clinical trial from 2015, Chilton et al. supposes positive effects on blood pressure, arterial stiffness and vascular resistance. So far there is no data about systemic vascular resistance and cardiac output in patients with type 2 diabetes with empagliflozin treatment or other SGLT2 inhibitors.
* Consequently, it remains currently unclear whether osmotic diuresis can be accounted for the longer term blood pressure lowering effects of empagliflozin, which remains stable also after new blood glucose equilibrium is reached.

ELIGIBILITY:
Inclusion Criteria:

1. Type 2 diabetes
2. Serum levels of HbA1c ≥ 6.5 %, despite treatment with diet and glucose lowering agents, which should include metformin (unless intolerance or contraindication to metformin exists)
3. Age ≥ 18 years
4. Participants of child-bearing age should use adequate contraception
5. Written informed consent prior to study participation

Exclusion Criteria:

1. Type 1 diabetes
2. Systolic blood pressure ≥ 160 mmHg, diastolic blood pressure ≥ 90 mmHg
3. Age ≥ 75 years
4. Pregnancy or lactating females
5. Urinary tract infections or significant formation of residual urine in medical history
6. Renal impairment (GFR < 30 ml/min/1.73 m2)
7. Liver disease (serum levels of AST, ALT or AP more than three times the upper limit of normal)
8. Uncontrolled thyroid disease
9. Endocrinopathies like Graves' disease, acromegaly, Cushing's disease
10. Hypertensive retinopathy or encephalopathy
11. Acute coronary syndrome, stroke or transient ischemic attack in last 6 weeks prior to randomization
12. The subject is mentally or legally incapacitated
13. The subject received an investigational drug within 30 days prior to inclusion into this study
14. Patients with newly diagnosed diabetes, who have not been subjected to diet and glucose lowering drug treatment.
15. Patients with particular risk for ketoacidosis (alcohol abuse, pancreatitis, pancreatic insulin deficiency from any cause, caloric restriction etc.) or ketoacidosis in the past
16. Frequent hypoglycaemic events (in the opinion of the investigator)
17. Patients in whom study participation is not deemed appropriate under consideration of clinical wellbeing by the principal investigator
18. Intolerance to Empagliflozin and excipients in Empagliflozin or rather placebo
19. Hypotension in the past (systolic blood pressure < 90 mmHg) in patients receiving treatment with blood lowering drugs
20. Signs of exsiccosis
21. Previous treatment with Empagliflozin in the past
22. Critically ill patients (in the opinion of the investigator)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2017-04-24 (Actual); Primary Completion 2019-01-23 (Actual); Study Completion 2019-01-23 (Actual)

PRIMARY OUTCOMES:
Mode of action | 3 months
  vascular resistance (dyn*s/cm^5)
Mode of action | 3 months
  cardiac output (l/min)

SECONDARY OUTCOMES:
Hemodynamics | 3 months
  Stroke volume (ml/beat)
Hemodynamics | 3 months
  stroke volume variation (%)
Energie expenditure | 3 months
  resting energy expenditure (calories/24h)
Cardio cascular | 3 months
  blood pressure (mmHg)
Urine | 3 months
  24 h sodium excretion (mmol/day)
Body weight | 3 months
  body weight (kg)
Cardio vascular | 3 months
  heart rate (bpm)
Blood | 3 months
  NT-proBNP (ng/l)
Blood | 3 months
  cystatin C(mg/dl)
Blood | 3 months
  serum levels of Glucose (mg/dl)
Blood | 3 months
  HbA1c (%)
Metabolism | 3 months
  total-ketone bodies (mmol/l)

CONTACTS AND LOCATIONS:
Overall Officials: Nikolaus Marx, Univ.-Prof. Dr. med., Principal Investigator — University Hospital, Aachen
Locations (1):
- Department of Internal Medicine I RWTH Aachen University Hospital, Aachen, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cherney DZ, Perkins BA, Soleymanlou N, Har R, Fagan N, Johansen OE, Woerle HJ, von Eynatten M, Broedl UC. The effect of empagliflozin on arterial stiffness and heart rate variability in subjects with uncomplicated type 1 diabetes mellitus. Cardiovasc Diabetol. 2014 Jan 29;13:28. doi: 10.1186/1475-2840-13-28. PMID 24475922
- [Background] Chilton R, Tikkanen I, Cannon CP, Crowe S, Woerle HJ, Broedl UC, Johansen OE. Effects of empagliflozin on blood pressure and markers of arterial stiffness and vascular resistance in patients with type 2 diabetes. Diabetes Obes Metab. 2015 Dec;17(12):1180-93. doi: 10.1111/dom.12572. Epub 2015 Oct 9. PMID 26343814
- [Background] DeFronzo RA, Hompesch M, Kasichayanula S, Liu X, Hong Y, Pfister M, Morrow LA, Leslie BR, Boulton DW, Ching A, LaCreta FP, Griffen SC. Characterization of renal glucose reabsorption in response to dapagliflozin in healthy subjects and subjects with type 2 diabetes. Diabetes Care. 2013 Oct;36(10):3169-76. doi: 10.2337/dc13-0387. Epub 2013 Jun 4. PMID 23735727
- [Background] Mauricio D. [Sodium-glucose co-transporter-2 inhibitors: from the bark of apple trees and familial renal glycosuria to the treatment of type 2 diabetes mellitus]. Med Clin (Barc). 2013 Sep;141 Suppl 2:31-5. doi: 10.1016/S0025-7753(13)70061-7. Spanish. PMID 24444522
- [Background] Sha S, Polidori D, Heise T, Natarajan J, Farrell K, Wang SS, Sica D, Rothenberg P, Plum-Morschel L. Effect of the sodium glucose co-transporter 2 inhibitor canagliflozin on plasma volume in patients with type 2 diabetes mellitus. Diabetes Obes Metab. 2014 Nov;16(11):1087-95. doi: 10.1111/dom.12322. Epub 2014 Jul 8. PMID 24939043
- [Background] Vasilakou D, Karagiannis T, Athanasiadou E, Mainou M, Liakos A, Bekiari E, Sarigianni M, Matthews DR, Tsapas A. Sodium-glucose cotransporter 2 inhibitors for type 2 diabetes: a systematic review and meta-analysis. Ann Intern Med. 2013 Aug 20;159(4):262-74. doi: 10.7326/0003-4819-159-4-201308200-00007. PMID 24026259
- [Background] Wanner C, Inzucchi SE, Lachin JM, Fitchett D, von Eynatten M, Mattheus M, Johansen OE, Woerle HJ, Broedl UC, Zinman B; EMPA-REG OUTCOME Investigators. Empagliflozin and Progression of Kidney Disease in Type 2 Diabetes. N Engl J Med. 2016 Jul 28;375(4):323-34. doi: 10.1056/NEJMoa1515920. Epub 2016 Jun 14. PMID 27299675
- [Background] Zinman B, Lachin JM, Inzucchi SE. Empagliflozin, Cardiovascular Outcomes, and Mortality in Type 2 Diabetes. N Engl J Med. 2016 Mar 17;374(11):1094. doi: 10.1056/NEJMc1600827. No abstract available. PMID 26981940